CLINICAL TRIAL: NCT04962542
Title: Comparison Between the Effect of Different Strategies of Ventilation During Cardiopulmonary Bypass on Arterial Oxygenation and Postoperative Pulmonary Dysfunction In Pediatric Patients With Congenital Non-cyanotic Heart Diseases
Brief Title: Ventilation During Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed sabry abdelsalam, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-74-2020
Record Dates: First submitted 2021-07-02; First posted 2021-07-15 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Lung Injury; Postoperative Complications; Pulmonary Collapse
MeSH Terms: conditions — Lung Injury; Postoperative Complications; Pulmonary Atelectasis | interventions — Ventilation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ventilated group (Active Comparator): the lungs will be kept inflated by delivery of oxygen : air 3 liter/min with FiO2 50% pressure-controlled mode, RR 20/min, PIP will be adjusted to keep Vt 2- 4 mL/kg as possible
  Interventions: Other: ventilation
- CPAP group (Active Comparator): lungs will be kept inflated by delivery of oxygen: air 3 liters/min with FiO2 50% and CPAP will be maintained via a circle system with airway pressure maintained at 5 cm H2O by PEEP valve
  Interventions: Other: ventilation
- controlled group (No Intervention): lungs will be deflated by disconnecting the breathing circuit from the ventilator (passive deflation).

INTERVENTIONS:
Other: ventilation — low volume positive pressure ventilation is better than continuous positive airway pressure and passive deflation on arterial oxygenation and PPD after CPB in pediatrics undergoing cardiac surgeries for non-cyanotic congenital heart defects.
  Arms: CPAP group; ventilated group

SUMMARY:
Postoperative pulmonary dysfunction (PPD) is a widely reported complication of cardiopulmonary bypass (CPB) although there is improvement in perioperative management, that leads to increased morbidity and mortality in cardiac surgery.

Many surgical-related factors can predispose to postoperative pulmonary complications such as the effects of general anesthesia combined with the effects of a median sternotomy, CPB, and the use of topical cooling for myocardial protection.

Main clinical manifestations of PPD include atelectasis, pleural effusion, and postoperative hypoxemia without clinical symptoms in addition to acute respiratory distress syndrome which is rare to happen but leads to high mortality Different strategies including perioperative management of mechanical ventilation (MV), restrictive transfusion, technical modifications of CPB, and medication administration such as steroids and aprotinin have been developed to lessen impairment of pulmonary function.

A recent meta-analysis identified improvement in oxygenation after weaning from CPB when low tidal volume (LTV) ventilation was maintained or after lung recruitment maneuvers (LRM), as compared to when there was no ventilation (noV). Also, maintaining mechanical ventilation may reduce the inflammation response and tissue damage. So far, available researches regarding whether ventilation during CPB could improve respiratory outcomes is still controversial especially in pediatric patients undergoing corrective surgeries for congenital heart defects.

DETAILED DESCRIPTION:
Our study is designed to determine the effect of different strategies of ventilation during CPB on arterial oxygenation and PPD in pediatrics undergoing corrective cardiac surgeries for non-cyanotic congenital anomalies.

Preoperative:

First, a proper and detailed history from the parents will be taken followed by a full and detailed examination of the child then the investigators will check all investigations including complete blood count(CBC), coagulation profile, liver enzymes, kidney function tests, chest X-ray (CXR), echocardiography, and blood grouping.

All patients will be premedicated with atropine 0.01 mg/kg, and midazolam 0.02 mg/kg intramuscular(IM), 30 minutes before induction of anesthesia.

Intraoperative:

the investigators will start with Standard Monitoring as ECG, Pulse oximetry, and non-invasive blood pressure. Then the investigators will proceed to induction using sevoflurane in 50% FiO2 followed by Placement of peripheral IV cannula and IV administration of fentanyl (2 µg/kg) and cisatracurium 0.1 mg/kg then Oral endotracheal intubation and the Capnogram will be connected to monitor End-tidal carbon dioxide(CO2).

The patient will be mechanically ventilated using pressure-controlled mode with a fraction of inspired oxygen(FiO2) 50%, Inspiration to expiration time ratio of 1:2, peak inspiratory pressure (PIP), and respiratory rate will be set according to the age to maintain the range of end-tidal carbon dioxide pressure at 35-45 mmHg in all groups.

Maintenance of anesthesia will be achieved using sevoflurane 2 % in 1:1 oxygen: air, cisatracurium infusion 1-2 mcg/kg/min and Fentanyl 1-5 µg/kg till the time of CPB (1 µg/kg before skin incision,2 µg/kg before sternotomy,2 µg/kg during cannulation) Advanced monitoring where nasopharyngeal temperature probe will be placed, a Central venous catheter to monitor central venous pressure(CVP), and Arterial cannula to monitor invasive blood pressure, then antibiotic will be given after skin test, Standard CPB technique will be used in all patients. Before aortic cannulation, patients will receive IV heparin 300-400 U.kg-1 aiming to produce activated clotting time (ACT) value > 400 sec. A membrane oxygenator (minimax plus; Medtronic's Inc., Anaheim, CA) will be used during CPB. Priming solution in the form of isotonic saline solution supplemented with heparin will be added to fresh whole blood in appropriate amounts to achieve a hematocrit of 20-25% during CPB. Furosemide in a dose of 1 mg/kg will be given to all patients. Anesthesia during CPB will be given by Sevoflurane administrated via a vaporizer inserted into the oxygenator gas supply with a constant gas flow of 3 liters/min. A non-pulsatile roller pump (model10.10.00; Stockett instruments; Munich, Germany) will be used and the pump flow will be adjusted at 2.4 to 2.6 L/min /m2 during the normothermic period targeting mean arterial blood pressure between 40 and 60 mmHg, Alpha-stat pH management was used and replacement fluids were added as blood (packed red cells), colloid or crystalloid as indicated.

After application of aortic cross-clamp, cold blood cardioplegia (20 mL/kg for initial dose) with 30 milliequivalent(mEq)/L of potassium, sodium bicarbonate 25 mEq/L, Xylocaine 120 mg/L will be injected into the aortic root, also topical myocardial cooling will be used.

During CPB the patients enrolled in the study will be randomly assigned to three groups using a computer-generated random sequence of numbers.

* Group A (n=20) the lungs will be kept inflated by delivery of oxygen: air 3 liters/min with FiO2 50% pressure-controlled mode, respiratory rate(RR) 20-30/min according to age, PIP will be adjusted to keep Vt 2 mL/kg as possible.
* Group B (n=20) their lungs will be kept inflated by delivery of oxygen: air 3 liters/min with FiO2 50% and continuous positive airway pressure(CPAP) will be maintained via a circle system with airway pressure maintained at 5 cmH2O by positive end expiratory pressure(PEEP) valve. This will be verified by a previously calibrated, in-circuit Bourdon gauge.
* Group C (control group) (n=20) their lungs will be deflated by disconnecting the breathing circuit from the ventilator (passive deflation).

Post CPB, the patient will be mechanically ventilated using pressure-controlled mode with FiO2 50%, Inspiration to expiration time ratio of 1:2, peak inspiratory pressure (PIP), and respiratory rate will be set according to the age to maintain the range of end-tidal carbon dioxide pressure at 35-45 mmHg in all groups.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologist(ASA) II, III.
* Patients with non-cyanotic congenital heart defects undergoing corrective surgeries during CPB [Atrial Septal Defect (ASD), Ventricular Septal Defect (VSD), Common A trio ventricular canal (CAVC)].

Exclusion Criteria:

* Any congenital anomalies of the lung as cystic fibrosis, congenial diaphragmatic hernia.

ASA IV. Patients with congenital cyanotic heart defects. Parents refusal.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
partial pressure of arterial oxygen(PaO2/FIO2) ratio 5 minutes after weaning from CPB. | 5 minutes after weaning from CPB
  measuring PaO2/FIO2 ratio in arterial blood gas sample

SECONDARY OUTCOMES:
PaO2/FIO2 ratio | after chest closure
  measuring PaO2/FIO2 ratio in arterial blood gas sample
PaO2/FIO2 ratio | 1 hour after arrival to ICU
  measuring PaO2/FIO2 ratio in arterial blood gas sample
Chest x-ray | 1 hour after arrival to ICU
  incidence of pleural effusion or lung collapse using portable x-ray machine
oxygenation index | 1 hour after arrival to ICU
  incidence of hypoxemic respiratory failure using an equation(fio2×mean airway pressure)/pao2

CONTACTS AND LOCATIONS:
Overall Officials: mohamed F yousef, MD, Study Director — professor of anesthesia. faculty of medicine. Cairo university
Locations (1):
- AbulReesh Hospital. faculty of medicine. cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided